CLINICAL TRIAL: NCT01700283
Title: Developing Objective Fatigue Indicators: Exploring the Relationships Among Fatigue, Muscle Power and Metabolomics Through Fatigue Management and Individualized Exercise Education Program in Colorectal Cancer Survivors.
Brief Title: Developing Objective Fatigue Indicators in Colorectal Cancer Survivors.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201208026RIC
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer、Fatigue、Muscle strength、Metabolomics
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exercise education and walking program (Experimental)
  Interventions: Behavioral: exercise education and walking program
- maintain their daily activity (No Intervention)

INTERVENTIONS:
Behavioral: exercise education and walking program — 12-week moderate intensity walking program
  Arms: exercise education and walking program

SUMMARY:
The aims of this four-year study are to

1. Explore exercise behavior, exercise barriers, and identify the significant factors for exercise behavior in colorectal cancer survivors.
2. Explore the relationships among fatigue, muscle strength, and metabolomics and further examine the possible biomarkers from muscle strength and metabolomics for fatigue.
3. Develop a clinical guidelines of home-based fatigue management and exercise program and test its effect on decreasing fatigue for patients with colorectal cancer after surgery in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer survivors completed treatment at least 3 months in clinics.
* Aged above 20.

Exclusion Criteria:

* KPS < 60
* Stage 4
* Bone meta

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Developing Objective Fatigue Indicators: Exploring the Relationships Among Fatigue, Muscle Power and Metabolomics Through Fatigue Management and Individualized Exercise Education Program in Colorectal Cancer Survivors | four-year study
  Develope the clinical exercise education program guideline for patients with early stage colorectal cancer survivor.

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ching Shun, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan